CLINICAL TRIAL: NCT04715295
Title: Open-label, Randomized Trial of the Safety and Efficacy of Doxycycline and Rivaroxaban Therapy Versus National Standard Therapy in Ambulatory Patients With Mild Symptomatic COVID-19
Brief Title: Safety and Efficacy of Doxycycline and Rivaroxaban in COVID-19
Acronym: DOXYCOV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yaounde Central Hospital (Other Government)
Responsible Party: Principal Investigator, Sobngwi Eugene, Medical Director, Yaounde Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNO0032020
Record Dates: First submitted 2020-10-02; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
Keywords: COVID-19; Doxycycline; Rivaroxaban; Hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Doxycycline; Rivaroxaban; Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycyclin and Rivaroxaban (Experimental): Oral Doxycyclin 200 mg daily for 7 days with or without Rivaroxaban
  Interventions: Drug: Doxycycline Tablets; Drug: Rivaroxaban 15Mg Tab
- National Standard (Active Comparator): Hydroxychloroquine 400 mg daily for 5 days in combination with Azithromycin 500 mg on day 1 and 250 mg daily from day 2 through day 5
  Interventions: Combination Product: Hydroxychloroquine and Azithromycin

INTERVENTIONS:
Drug: Doxycycline Tablets — Doxycycline 200 mg daily for 7 days
  Other Names: Doxycycline
  Arms: Doxycyclin and Rivaroxaban
Drug: Rivaroxaban 15Mg Tab — Rivaroxaban 15 mg tablets daily from day 1 to day 10
  Arms: Doxycyclin and Rivaroxaban
Combination Product: Hydroxychloroquine and Azithromycin — Hydroxychloroquine 400mg daily from day 1 to day 5 in combination with Azithromycin 500mg on day 1 and 250 mg daily from day 2 to day 5
  Arms: National Standard

SUMMARY:
This is an exploratory study to evaluate the efficacy of Doxycycline (200mg on D1 to D7) and Rivaroxaban (15 mg daily on D1 to D7) versus the combination of Hydroxychloroquine (400 mg on D1 to D7) and Azithromycin (500 mg on D1 and 250mg on D2 to D5) as per national standard to treat ambulatory mild COVID-19 patients, with the aim to achieve early negativity of RT-PCR of SARS-CoV-2 from nasopharyngeal swab, and early clinical improvement and prevention of severe disease.

DETAILED DESCRIPTION:
This is an exploratory study to evaluate the efficacy of Doxycycline (200mg on D1 to D7) and Rivaroxaban (15 mg on D1 to D7) versus combination of hydroxychloroquine (400 mg on D1 to D7) and azithromycin (500 mg on D1 and 250mg on D2 to D5) to treat ambulatory patients with mild COVID-19.

We aim to demonstrate early improvement of a clinical core set of outcomes and prevention of clinical worsening, and early negativity of SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) among ambulatory patients with mild COVID-19 by treating them with Doxycycline and Rivaroxaban compared to patients who receive Hydroxychloroquine and Azithromycin as per National standard therapy of COVid-19.

Ambulatory patients with mild symptoms and with confirmed diagnosis of COVID-19 will receive the treatment.

The primary objective of the study is to evaluate the Safety and Efficacy of Doxycycline and Rivaroxaban versus National standard therapy of mild COVid-19.

The primary endpoint is failure (i.e severe evolution) measured as PaO2 < 92% within 10 days after initiation of treatment.

The secondary objectives of the study are to evaluate

* Safety of the different investigational therapies up to D10 days of follow-up per arm,
* Hospitalisation due to Covid 19 infection rate per arm,
* Time to hospitalisation due to Covid 19 infection,
* Cure rate by treatment arm and Death rate,
* Worsening as assessed by the need for additional concomitant medication,
* Efficacy in sub-groups of patients (with pre-existing conditions/co-morbidities and by age group).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection confirmed by SARS-Cov2 - RT PCR - as per protocol
* Able to start the treatment within 24 hours from time of diagnosis
* Patient with mild symptoms as defined by WHO, with PaO2 > 93%
* Signed written consent of the patient
* Accepts and has the ability to be reached by phone during the study duration, plus a designated a contact person who can be contacted in case of emergency

Exclusion Criteria:

* Blood pressure < 90/60mm Hg
* Respiratory rate ≥ 30/min
* Known cardiac condition
* Known G6PD deficiency
* Patients with < 45kg
* eGFR < 30 ml/min or ALT ≥ 3N or body temperature ≥ 38°C or any life-threatening comorbidity
* Any reason that makes it impossible to monitor the patient during the study period
* Baseline ECG prior to randomization showing QTc > 500 ms
* Ongoing treatment other than symptomatic
* history of retinopathy
* Absolute contra-indication to treatment with hydroxychloroquine (known hypersensitivity, concomitant treatment at risk of torsades de pointes)
* Contraindication to any study medication including allergy
* Ongoing treatment with high dose systemic chronic corticosteroid (> 40 mg)
* Patients treated by immunosuppressants treatment at the time of randomization
* Known Pregnant women and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-09-05 (Estimated)

PRIMARY OUTCOMES:
Clinical | Day 1 to 10
  Change of Clinical stage of COVID-19
Virological | Day 1 to 10
  Time to negativity of SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) on nasopharyngeal swab.

SECONDARY OUTCOMES:
Symptom remission | Day 1 to 10
  Time to remission of symptoms in days
Hospitalisation | Day 1 to 10
  Need for hospitalisation due to worsening
Mortality | Day 1 to 10
  All-cause mortality
Biological variables | Day 1 to Day 7 and Day 10
  Change from baseline of WBC count

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Sobngwi, Principal Investigator — University of Yaounde 1
Locations (1):
- Yaounde Central Hospital, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request and approval by the National COVID19 Scientific Board
Supporting Information: Study Protocol, SAP, CSR
Time Frame: one year after completion
Access Criteria: Data will be shared upon request and approval by the National COVID19 Scientific Board

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523